CLINICAL TRIAL: NCT07173959
Title: Digital Therapy for Individualized Intervention and Management of Gestational Diabetes Mellitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: K8156
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Gestational Diabetes Mellitus (GDM)
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): This group of pregnant women received nutritional intervention and feedback provided by a digital therapy product (mini-program) relying on an AI system on the basis of routine obstetric care
  Interventions: Device: GDM digital Therapy mini-program
- control group (Placebo Comparator): Pregnant women randomly assigned to the control group used a mini-program that looked the same as digital therapy products but only had educational and recording functions on the basis of routine obstetric care
  Interventions: Device: Pregnancy record and education mini-program

INTERVENTIONS:
Device: GDM digital Therapy mini-program — The main functions of digital therapy products include personalized recipe recommendations, exercise and diet records and personalized analysis, blood sugar and weight monitoring, and the generation of weekly and monthly electronic comprehensive reports. The content of the electronic comprehensive reports includes the weight gain, blood sugar status, examination indicators, mood, and the proportion of diet and exercise of pregnant women in line with the system's recommendations during this period of time.
  Arms: intervention group
Device: Pregnancy record and education mini-program — This mini-program looks the same as digital therapy products but only has the functions of education and record-keeping
  Arms: control group

SUMMARY:
Existing studies have shown that the management combined with digital health technology can increase the qualified rate of blood glucose in pregnant women with gestational diabetes mellitus (GDM), and the earlier the intervention, the better the effect of blood glucose control. Previously, there was a lack of relevant research on digital therapeutics for the systematic management of gestational diabetes in China. A data-driven digital therapy product for gestational diabetes (doctor's end + patient's end) was established. This product integrates functions such as information recording, risk assessment, evaluation and suggestion, prescription issuance, and knowledge popularization. It aims to provide personalized blood glucose regulation plans for pregnant women with gestational diabetes and enhance the health awareness and self-management ability of families with gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 24 to 28 weeks of pregnancy GDM was diagnosed by OGTT test single pregnancy Be able to use smart phone APP to conduct intervention management based on digital therapy software program

Exclusion Criteria:

* Suffering from type 1 or type 2 diabetes Other serious organic diseases With severe mental disorders Intervention management cannot be carried out as planned using digital therapeutics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of achieving blood glucose targets | From enrollment to the end of treatment at 16 weeks

SECONDARY OUTCOMES:
Weight gain during pregnancy | From enrollment to the end of treatment at 16 weeks
The incidence of adverse pregnancy outcomes | During childbirth

IPD SHARING:
Plan to Share IPD: No